CLINICAL TRIAL: NCT04114292
Title: A Phase I Open Label Study of the Efficacy and Safety of Tudca in Ulcerative Colitis
Brief Title: TUDCA as a Therapy for Ulcerative Colitis (UC)
Acronym: TUDCA
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Washington University School of Medicine (Other)
Collaborators: Crohn's and Colitis Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 201812101
Record Dates: First submitted 2019-09-25; First posted 2019-10-03 (Actual); Last update posted 2021-12-22 (Actual); Status verified 2021-12

CONDITIONS: Ulcerative Colitis
Keywords: Ulcerative Colitis; tudca; tauroursodeoxycholic acid
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Intervention Model Description: Determine the effect of TUDCA treatment on colon inflammation including ER stress in colon biopsy tissues from subjects with symptomatic ulcerative colitis. Secondary: Measure the safety, tolerance and efficacy of TUDCA treatment in symptomatic ulcerative colitis.
Masking Description: Open-label study. All patients will receive TUDCA.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- TUDCA (Experimental): 1.75-2 grams daily in divided dosing
  Interventions: Drug: Tauroursoursodeoxycholic acid, brand name Tudcabil

INTERVENTIONS:
Drug: Tauroursoursodeoxycholic acid, brand name Tudcabil — Dosed in capsules containing 250 or 500mg of TUDCA for a total dose of 1.75-2g/day
  Other Names: Tudcabil

SUMMARY:
This is a Phase I open label study examining the efficacy and safety of TUDCA (tauroursodeoxycholic acid) in ulcerative colitis treatment.

DETAILED DESCRIPTION:
TUDCA (tauroursodeoxycholic acid) is a dietary supplement that has shown to reduce cellular stress related to inflammation. In this Phase I study, patients with active ulcerative colitis will be receive TUDCA for six weeks. Safety and tolerability will be assessed. Efficacy will be assessed using ulcerative colitis disease activity measurements as well as markers of intestinal inflammation before and after treatment. The overall goal of this project is to determine TUDCA can provide a new therapeutic option with a desirable safety profile for patients with ulcerative colitis focused on the inflamed intestinal epithelium.

ELIGIBILITY:
Inclusion Criteria:

* Ages Eligible for Study: 18 Years to 65 Years;
* Confirmed ulcerative colitis disease through radiographic, endoscopic and/or histologic criteria;
* Confirmed with active ulcerative colitis (defined as a complete Mayo score ≥ 5 with endoscopic subscore of ≥ 1) See Appendix for Mayo Score using recent adaptation to include any friability on endoscopy to be scored as "2".
* On a stable dose of medications for inflammatory bowel disease (IBD) (i.e. no change in medication within 4 weeks of study enrollment) and not planning to initiate new medication other than TUDCA.

Exclusion Criteria:

* Those that received other chemical chaperone therapies in the 3 months prior to screening;
* Individuals accompanied by gallstones, other intestinal disorders or cancers, or any possible cholestatic pathologies that could alter the enterohepatic circulation of the bile acids, including previous cholecystectomy or short bowel syndrome;
* Subjects with alcohol or drug abuse within the recent year;
* Serious heart, lung, kidney, digestive, nervous, mental, or autoimmune diseases
* Those with plans for abdominal surgery;
* Those unable or unwilling to provide informed consent or failure to comply with the test requirements;
* Pregnant, lactating women;
* Those receiving or planning to receive medicines that inhibit the absorption of the bile acids in the intestine;
* All female subjects must have birth control and not plan to become pregnant during the study. As TUDCA may interfere in the absorption of oral contraceptives, the acceptable methods of birth control should include abstinence or 2 of the following intrauterine device (IUD-with or without local hormone release), diaphragm, spermicides, cervical cap, contraceptive sponge, and /or condoms.
* Subjects with baseline liver transamines (AST or ALT) > 1.5 X the upper limit of normal.
* Patients with complete biliary obstruction and known hypersensitivity or intolerance to TUDCA or any of the components of Tudcabil (or to other bile acids).
* Patients with moderate-to-severe hepatic impairment.
* Evidence of worsening liver function based on the 2 initial laboratory values used to establish the baseline.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Estimated)
Dates: Start 2019-01-17 (Actual); Primary Completion 2022-07-31 (Estimated); Study Completion 2022-07-31 (Estimated)

PRIMARY OUTCOMES:
Determine the effect of TUDCA treatment on ER stress in colon biopsy tissues from subjects with symptomatic ulcerative colitis | Baseline and post 6 weeks of TUDCA treatment
  Change in ER stress markers as measured by expression of X box binding protein-1 (XBP1), Binding immunoglobulin protein (BIP) and Eukaryotic Translation Initiation Factor 2A (eIF2a) in colon biopsy tissues before and after 6 weeks of TUDCA treatment.

SECONDARY OUTCOMES:
Monitoring of UC patients for TUDCA safety and tolerability: Adverse events | Every 2 weeks after starting TUDCA until 2 weeks after completing 6 weeks of TUDCA treatment. (i.e. study points weeks 2, 4, 6 and 8)
  Monitor and define TUDCA safety/tolerability in this population through frequent monitoring and symptom assessment as detailed in the study procedures. Adverse events will be categorized according to CTCAE v5.0 criteria and grading.
Change ulcerative colitis disease activity based on Total Mayo Score | Baseline and post 6 weeks of TUDCA treatment
  The Mayo Ulcerative colitis score is an aggregate of individual parameters evaluating rectal bleeding, stool frequency, endoscopic severity and physicians global assessment. Each of these subscores has a range from 0-3 where 3 is worse. a total score can range from 0 to 12 with 0 being in remission and 12 representing the most severe disease. As this is a secondary endpoint in a small trial, patients total scores (out of 12) will be compared from baseline to week 6 using a paired students t test. Mayo score reference is Schroeder KW, Tremaine WJ, Ilstrup DM. Coated oral 5-aminosalicylic acid therapy for mildly to moderately active ulcerative colitis. A randomized study. N Engl J Med 1987;317:1625-9.
Change in inflammation on histology by Goebes index | Baseline and post 6 weeks of TUDCA treatment
  The Geboes histology index is a reproducible grading scale for histological assessment of inflammation in ulcerative colitis. This is a six grade classification system for inflammation which can also be fine tuned within each grade. The grades are: 0, structural change only; 1, chronic inflammation; 2, lamina propria neutrophils; 3, neutrophils in epithelium; 4, crypt destruction; and 5, erosions or ulcers. As this is a secondary endpoint in a small trial, patients total scores (out of 20) will be compared from baseline to week 6 using a paired students t test. Higher scores represent more severe disease. The reference for the Geboes index is "Geboes K, Riddell R, Ost A, et al. A reproducible grading scale for histological assessment of inflammation in ulcerative colitis. Gut 2000;47:404-9."

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Barnes-Jewish West County Hospital, Creve Coeur, Missouri
  - Barnes-Jewish Hospital, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kaser A, Lee AH, Franke A, Glickman JN, Zeissig S, Tilg H, Nieuwenhuis EE, Higgins DE, Schreiber S, Glimcher LH, Blumberg RS. XBP1 links ER stress to intestinal inflammation and confers genetic risk for human inflammatory bowel disease. Cell. 2008 Sep 5;134(5):743-56. doi: 10.1016/j.cell.2008.07.021. PMID 18775308
- [Background] Adolph TE, Tomczak MF, Niederreiter L, Ko HJ, Bock J, Martinez-Naves E, Glickman JN, Tschurtschenthaler M, Hartwig J, Hosomi S, Flak MB, Cusick JL, Kohno K, Iwawaki T, Billmann-Born S, Raine T, Bharti R, Lucius R, Kweon MN, Marciniak SJ, Choi A, Hagen SJ, Schreiber S, Rosenstiel P, Kaser A, Blumberg RS. Paneth cells as a site of origin for intestinal inflammation. Nature. 2013 Nov 14;503(7475):272-6. doi: 10.1038/nature12599. Epub 2013 Oct 2. PMID 24089213
- [Background] Cao SS, Song B, Kaufman RJ. PKR protects colonic epithelium against colitis through the unfolded protein response and prosurvival signaling. Inflamm Bowel Dis. 2012 Sep;18(9):1735-42. doi: 10.1002/ibd.22878. Epub 2012 Jan 24. PMID 22275310
- [Background] Cao SS, Zimmermann EM, Chuang BM, Song B, Nwokoye A, Wilkinson JE, Eaton KA, Kaufman RJ. The unfolded protein response and chemical chaperones reduce protein misfolding and colitis in mice. Gastroenterology. 2013 May;144(5):989-1000.e6. doi: 10.1053/j.gastro.2013.01.023. Epub 2013 Jan 18. PMID 23336977
- [Background] Cao SS, Wang M, Harrington JC, Chuang BM, Eckmann L, Kaufman RJ. Phosphorylation of eIF2alpha is dispensable for differentiation but required at a posttranscriptional level for paneth cell function and intestinal homeostasis in mice. Inflamm Bowel Dis. 2014 Apr;20(4):712-22. doi: 10.1097/MIB.0000000000000010. PMID 24577114
- [Background] Wang S, Kaufman RJ. The impact of the unfolded protein response on human disease. J Cell Biol. 2012 Jun 25;197(7):857-67. doi: 10.1083/jcb.201110131. PMID 22733998
- [Background] Shkoda A, Ruiz PA, Daniel H, Kim SC, Rogler G, Sartor RB, Haller D. Interleukin-10 blocked endoplasmic reticulum stress in intestinal epithelial cells: impact on chronic inflammation. Gastroenterology. 2007 Jan;132(1):190-207. doi: 10.1053/j.gastro.2006.10.030. Epub 2006 Oct 21. PMID 17241871
- [Background] Hu S, Ciancio MJ, Lahav M, Fujiya M, Lichtenstein L, Anant S, Musch MW, Chang EB. Translational inhibition of colonic epithelial heat shock proteins by IFN-gamma and TNF-alpha in intestinal inflammation. Gastroenterology. 2007 Dec;133(6):1893-904. doi: 10.1053/j.gastro.2007.09.026. Epub 2007 Sep 25. PMID 18054561
- [Background] Heazlewood CK, Cook MC, Eri R, Price GR, Tauro SB, Taupin D, Thornton DJ, Png CW, Crockford TL, Cornall RJ, Adams R, Kato M, Nelms KA, Hong NA, Florin TH, Goodnow CC, McGuckin MA. Aberrant mucin assembly in mice causes endoplasmic reticulum stress and spontaneous inflammation resembling ulcerative colitis. PLoS Med. 2008 Mar 4;5(3):e54. doi: 10.1371/journal.pmed.0050054. PMID 18318598
- [Background] McGovern DP, Gardet A, Torkvist L, Goyette P, Essers J, Taylor KD, Neale BM, Ong RT, Lagace C, Li C, Green T, Stevens CR, Beauchamp C, Fleshner PR, Carlson M, D'Amato M, Halfvarson J, Hibberd ML, Lordal M, Padyukov L, Andriulli A, Colombo E, Latiano A, Palmieri O, Bernard EJ, Deslandres C, Hommes DW, de Jong DJ, Stokkers PC, Weersma RK; NIDDK IBD Genetics Consortium; Sharma Y, Silverberg MS, Cho JH, Wu J, Roeder K, Brant SR, Schumm LP, Duerr RH, Dubinsky MC, Glazer NL, Haritunians T, Ippoliti A, Melmed GY, Siscovick DS, Vasiliauskas EA, Targan SR, Annese V, Wijmenga C, Pettersson S, Rotter JI, Xavier RJ, Daly MJ, Rioux JD, Seielstad M. Genome-wide association identifies multiple ulcerative colitis susceptibility loci. Nat Genet. 2010 Apr;42(4):332-7. doi: 10.1038/ng.549. Epub 2010 Mar 14. PMID 20228799
- [Derived] Lamm V, Huang K, Deng R, Cao S, Wang M, Soleymanjahi S, Promlek T, Rodgers R, Davis D, Nix D, Escudero GO, Xie Y, Chen CH, Gremida A, Rood RP, Liu TC, Baldridge MT, Deepak P, Davidson NO, Kaufman RJ, Ciorba MA. Tauroursodeoxycholic Acid (TUDCA) Reduces ER Stress and Lessens Disease Activity in Ulcerative Colitis. medRxiv [Preprint]. 2025 Apr 4:2025.04.02.25322684. doi: 10.1101/2025.04.02.25322684. PMID 40236400

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-11): https://cdn.clinicaltrials.gov/large-docs/92/NCT04114292/Prot_SAP_000.pdf